CLINICAL TRIAL: NCT00180986
Title: Randomized Trial Of Platelet Transfusion Policies After Blood Stem Cells Transplantation In Young Children: Reduction Of Number Of Single Platelet Concentrate Donors Per Child
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Minnie; CSET 94/357
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2005-12-14 (Estimated); Status verified 2005-09

CONDITIONS: Children Treated With High-Dose Chemotherapy (HDC) Followed by Haematopoietic Stem Cell Transplantation (HSCT)

INTERVENTIONS:
Procedure: Platelet concentrates

SUMMARY:
Randomized Trial Of Platelet Transfusion Policies After Blood Stem Cells Transplantation In Young Children: Reduction Of Number Of Single Platelet Concentrate Donors Per Child

ELIGIBILITY:
Inclusion Criteria:

* Children weighing 30 kg or less with a diagnosis of haematological malignancy or solid tumour, who were candidates for HSCT were eligible for inclusion in the study.
* Written informed consent was required from parents of eligible children.

Exclusion Criteria:

* Children were excluded if they had a anti-HLA and/or anti-HPA antibody, if they were prior included in this study or if the parents declined to participate.

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120
Dates: Start 1995-10

PRIMARY OUTCOMES:
The primary end point of the study was tocompare the number of platelet concentrates donors who were implicated in platelet transfusion supportive after HSCT.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie LAPIERRE, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave-Roussy, Villejuif, France